CLINICAL TRIAL: NCT00056771
Title: Clinical and Molecular Studies in Families With Congenital or Hereditary Cataracts
Brief Title: Clinical and Genetic Studies of Families With Congenital or Hereditary Cataracts
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030123; 03-EI-0123
Record Dates: First submitted 2003-03-22; First posted 2003-03-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-05-25

CONDITIONS: Cataract
Keywords: Cataract; Congenital Cataracts; Hereditary Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will explore the clinical and hereditary (genetic) features of inherited cataracts. A cataract is a clouding of the eye lens, which focuses light on the back of the eye. When the lens becomes cloudy and does not let light through, vision is impaired. Cataracts may be associated with vision problems alone, or with other problems, such as changes in facial appearance or skin problems. A better understanding of these genetic conditions may help in the development of better diagnostic tests.

Patients with inherited cataracts and their family members may be eligible for this study. Participants will be drawn from patients enrolled in other studies of inherited cataracts at the NEI and collaborating clinics.

Participants will undergo the following tests and procedures:

* Medical and surgical history;
* Verification of diagnosis;
* Construction of a family tree regarding familial vision problems;
* Complete eye examination, including dilation of the pupils and photography of the lens, tests of color vision and field of vision, and of the ability to see in the dark;
* Blood sample collection (20 ml, or 4 teaspoons) for genetic studies of hereditary cataracts.

DETAILED DESCRIPTION:
Objective: This project, Clinical and Molecular Studies in Families with Congenital or Hereditary Cataracts will study the inheritance of genetic cataracts, both Mendelian and complex age related cataracts, in families of many nationalities and ethnic backgrounds in order to identify the genes that, when mutated, cause cataracts and the pathophysiology through which they act.

Study Population: Families of many nationalities and ethnic backgrounds. We will study a maximum or 5,000 patients and family members.

Design: The study consists of ascertaining individuals, and especially families with multiple individuals, affected by both congenital and age related cataracts. These patients and their families will undergo detailed ophthalmological examinations to characterize their cataracts and determine their affectation status. A blood sample will be collected from each individual for isolation of DNA and in some individuals for lymphoblastoid transformation to establish a renewable source of DNA. Linkage analysis, physical mapping, and mutational screening will be carried out to identify the specific the gene and the mutations in it that are associated with cataracts in this family. If necessary, the gene product will be characterized biochemically. The study will enroll subjects at NEI and collaborating institutions, the Centre for Excellence in Molecular Biology, Lahore, Pakistan, the Zhongshan Ophthalmic Center, Guangzhou, China, the Aravind Eye Hospital, Madurai, India, and the University of Parma, Italy and the All India Institute of Medical Sciences (AIIMS).

Outcome Measures: Linkage will be determined using the lod score method and mutations in specific genes will be assessed using a combination of residue conservation, blosum score, and molecular modeling. Biochemical, metabolic, and physiological effects will be individualized to the specific assay.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with the following will be recruited:

1. Individuals or family members of individuals with inherited cataracts, either congenital, childhood, or age related.
2. Adults must be capable of providing their own consent.
3. All subjects must be able to cooperate with study examination and phlebotomy.
4. Older than 4 years of age.

EXCLUSION CRITERIA:

1. Diseases, infections, or trauma that mimic inherited cataracts.
2. Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3432 (Actual)
Dates: Start 2003-03-18; Study Completion 2016-05-25

PRIMARY OUTCOMES:
statistically significant linkage

CONTACTS AND LOCATIONS:
Overall Officials: James F Hejtmancik, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (5):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Zhongshan Ophthalmic Center, Guangzhou, China
- Aravind Eye Hospital, Maduri, India
- University of Parma, Parma, Italy
- Centre for Excellence in Molecular Biology, Lahore, Pakistan

REFERENCES:
- [Background] Ostrovsky MA, Sergeev YV, Atkinson DB, Soustov LV, Hejtmancik JF. Comparison of ultraviolet induced photo-kinetics for lens-derived and recombinant beta-crystallins. Mol Vis. 2002 Mar 20;8:72-8. PMID 11951082
- [Background] Sheets NL, Chauhan BK, Wawrousek E, Hejtmancik JF, Cvekl A, Kantorow M. Cataract- and lens-specific upregulation of ARK receptor tyrosine kinase in Emory mouse cataract. Invest Ophthalmol Vis Sci. 2002 Jun;43(6):1870-5. PMID 12036992
- [Background] Chen WV, Fielding Hejtmancik J, Piatigorsky J, Duncan MK. The mouse beta B1-crystallin promoter: strict regulation of lens fiber cell specificity. Biochim Biophys Acta. 2001 May 28;1519(1-2):30-8. doi: 10.1016/s0167-4781(01)00201-9. PMID 11406268